CLINICAL TRIAL: NCT00043836
Title: A Pilot Study Of ALT-711 In Elderly Patients With Isolated Diastolic Heart Failure: The DIAMOND Study
Brief Title: The DIAMOND Study: Distensibility Improvement And Remodeling in Diastolic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synvista Therapeutics, Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALT-711-0214
Record Dates: First submitted 2002-08-14; First posted 2002-08-15 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2007-08

CONDITIONS: Heart Failure, Congestive; Dyspnea; Pulmonary Edema
Keywords: ejection fraction; exercise tolerance; heart failure, congestive; quality of life
MeSH Terms: conditions — Heart Failure; Dyspnea; Pulmonary Edema | interventions — alagebrium

INTERVENTIONS:
Drug: ALT-711

SUMMARY:
The purpose of this study is to test the hypothesis that treatment with oral ALT-711 twice daily for 16 weeks will improve aortic distensibility, exercise tolerance, and quality of life in elderly patients with isolated diastolic heart failure (DHF), and that the improvements in exercise tolerance will correlate with the improvements in aortic distensibility.

ELIGIBILITY:
Inclusion Criteria

1. Men or women ≥ 60 years of age.
2. Diagnosis of congestive heart failure with one or both of the following criteria: a Heart Failure Clinical Score ≥ 3 based on the NHANES-I criteria and/or a history of either acute pulmonary edema or the occurrence of 2 or more of the following with subsequent improvement with diuretic therapy and with no other identifiable cause: dyspnea on exertion, paroxysmal nocturnal dyspnea, orthopnea, systemic edema, exertional fatigue.
3. Left ventricular ejection fraction ≥ 50% based on the baseline Doppler echocardiography test.
4. Ability to provide written informed consent.
5. Ability to comply with procedures specified in the study protocol.

Exclusion Criteria

1. Valvular heart disease as the primary etiology of congestive heart failure.
2. Significant change in cardiovascular medication(s) <3 weeks prior to the baseline visit.
3. Uncontrolled hypertension.
4. History of stroke, or any sequelae of a transient ischemic attack (TIA), reversible ischemic neurologic defect (RIND), or stroke, within the last 12 months prior to entry into the study.
5. Cancer or other noncardiovascular conditions with life expectancy less than 2 years.
6. Significant anemia defined as a hemoglobin <11 gm/dL.
7. Significant renal insufficiency defined as a serum creatinine >2.5 mg/dL.
8. Significant hepatic insufficiency defined as an SGPT (ALT) or SGOT (AST) >2.5 times the upper limit of normal.
9. Psychiatric disease (including uncontrolled major psychoses, depression, dementia, or personality disorder) or any additional condition(s) which, in the investigator's opinion, would prohibit the patient from completing the study, or not be in the best interest of the patient.
10. Presence or history of drug or alcohol abuse.
11. Prior exposure to ALT-711 or use of any other investigational drugs within 30 days prior to screening.
12. Known seropositivity for HIV or hepatitis C, or presence of hepatitis B surface antigen.
13. Severe COPD requiring recurrent oral steroids, oxygen at home or more than one inhaler.
14. Baseline echocardiogram demonstrating the presence of left ventricular ejection fraction <50%.
15. Unstable or uncontrolled myocardial ischemia, with no wall abnormality.
16. Screening Familiarization Exercise Test demonstrating the presence of any of the following findings: evidence of significant ischemia (consisting of ECG finding of > 1 mm flat ST depression confirmed with echocardiogram wall motion, or wall motion abnormality or decrease in global contractility on echocardiogram, or inability to continue exercising due to significant chest or leg pain or any reason other than exhaustion/fatigue/dyspnea, exercise SBP >240 mm Hg, DBP >110 mmHg, unstable hemodynamics or rhythm, or unwilling or unable to complete test adequately.
17. Any contraindications to magnetic resonance imaging including but not limited to indwelling metal-containing prosthesis (orthopedic, valvular, other), pacemaker or defibrillator, history of welding occupation (ocular metal debris), or uncontrollable claustrophobia.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2002-07; Primary Completion 2003-02 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W Kitzman, MD, Principal Investigator — Associate Professor of Medicine and Cardiology, Wake Forest University Baptist Medical Center; Michael R Zile, MD, Principal Investigator — Charles Ezra Daniel Professor of Medicine, Medical University of South Carolina
Locations (2):
- United States (2):
  - Wake Forest University Baptist Medical Center, Department of Cardiology, Winston-Salem, North Carolina
  - Medical University of South Carolina and Ralph H. Johnson VA Medical Center, Charleston, South Carolina

REFERENCES:
- [Background] Asif M, Egan J, Vasan S, Jyothirmayi GN, Masurekar MR, Lopez S, Williams C, Torres RL, Wagle D, Ulrich P, Cerami A, Brines M, Regan TJ. An advanced glycation endproduct cross-link breaker can reverse age-related increases in myocardial stiffness. Proc Natl Acad Sci U S A. 2000 Mar 14;97(6):2809-13. doi: 10.1073/pnas.040558497. PMID 10706607
- [Background] Hundley WG, Kitzman DW, Morgan TM, Hamilton CA, Darty SN, Stewart KP, Herrington DM, Link KM, Little WC. Cardiac cycle-dependent changes in aortic area and distensibility are reduced in older patients with isolated diastolic heart failure and correlate with exercise intolerance. J Am Coll Cardiol. 2001 Sep;38(3):796-802. doi: 10.1016/s0735-1097(01)01447-4. PMID 11527636
- [Background] Kass DA, Shapiro EP, Kawaguchi M, Capriotti AR, Scuteri A, deGroof RC, Lakatta EG. Improved arterial compliance by a novel advanced glycation end-product crosslink breaker. Circulation. 2001 Sep 25;104(13):1464-70. doi: 10.1161/hc3801.097806. PMID 11571237
- [Background] Kitzman DW, Gardin JM, Gottdiener JS, Arnold A, Boineau R, Aurigemma G, Marino EK, Lyles M, Cushman M, Enright PL; Cardiovascular Health Study Research Group. Importance of heart failure with preserved systolic function in patients > or = 65 years of age. CHS Research Group. Cardiovascular Health Study. Am J Cardiol. 2001 Feb 15;87(4):413-9. doi: 10.1016/s0002-9149(00)01393-x. PMID 11179524
- [Background] Kitzman DW. Heart Failure in the Elderly: Systolic and Diastolic Dysfunction. Am J Geriatr Cardiol. 1996 Jan;5(1):20-26. No abstract available. PMID 11416361
- [Background] Little WC, Ohno M, Kitzman DW, Thomas JD, Cheng CP. Determination of left ventricular chamber stiffness from the time for deceleration of early left ventricular filling. Circulation. 1995 Oct 1;92(7):1933-9. doi: 10.1161/01.cir.92.7.1933. PMID 7671378
- [Background] Marburger CT, Brubaker PH, Pollock WE, Morgan TM, Kitzman DW. Reproducibility of cardiopulmonary exercise testing in elderly patients with congestive heart failure. Am J Cardiol. 1998 Oct 1;82(7):905-9. doi: 10.1016/s0002-9149(98)00502-5. PMID 9781977
- [Background] Vaitkevicius PV, Lane M, Spurgeon H, Ingram DK, Roth GS, Egan JJ, Vasan S, Wagle DR, Ulrich P, Brines M, Wuerth JP, Cerami A, Lakatta EG. A cross-link breaker has sustained effects on arterial and ventricular properties in older rhesus monkeys. Proc Natl Acad Sci U S A. 2001 Jan 30;98(3):1171-5. doi: 10.1073/pnas.98.3.1171. PMID 11158613
- [Background] Warner JG Jr, Metzger DC, Kitzman DW, Wesley DJ, Little WC. Losartan improves exercise tolerance in patients with diastolic dysfunction and a hypertensive response to exercise. J Am Coll Cardiol. 1999 May;33(6):1567-72. doi: 10.1016/s0735-1097(99)00048-0. PMID 10334425
- [Background] Wolffenbuttel BH, Boulanger CM, Crijns FR, Huijberts MS, Poitevin P, Swennen GN, Vasan S, Egan JJ, Ulrich P, Cerami A, Levy BI. Breakers of advanced glycation end products restore large artery properties in experimental diabetes. Proc Natl Acad Sci U S A. 1998 Apr 14;95(8):4630-4. doi: 10.1073/pnas.95.8.4630. PMID 9539789
- [Background] Zile MR, Brutsaert DL. New concepts in diastolic dysfunction and diastolic heart failure: Part I: diagnosis, prognosis, and measurements of diastolic function. Circulation. 2002 Mar 19;105(11):1387-93. doi: 10.1161/hc1102.105289. No abstract available. PMID 11901053
- [Background] Zile MR, Brutsaert DL. New concepts in diastolic dysfunction and diastolic heart failure: Part II: causal mechanisms and treatment. Circulation. 2002 Mar 26;105(12):1503-8. doi: 10.1161/hc1202.105290. No abstract available. PMID 11914262
- [Background] Zile MR, Gaasch WH, Carroll JD, Feldman MD, Aurigemma GP, Schaer GL, Ghali JK, Liebson PR. Heart failure with a normal ejection fraction: is measurement of diastolic function necessary to make the diagnosis of diastolic heart failure? Circulation. 2001 Aug 14;104(7):779-82. doi: 10.1161/hc3201.094226. PMID 11502702
- [Background] Kitzman DW. Diastolic heart failure in the elderly. Heart Fail Rev. 2002 Jan;7(1):17-27. doi: 10.1023/a:1013745705318. PMID 11790920
- [Background] Kitzman DW. Heart failure with normal systolic function. Clin Geriatr Med. 2000 Aug;16(3):489-512. doi: 10.1016/s0749-0690(05)70025-2. PMID 10918644
- [Background] Kitzman DW. Diastolic dysfunction in the elderly. Genesis and diagnostic and therapeutic implications. Cardiol Clin. 2000 Aug;18(3):597-617, x. doi: 10.1016/s0733-8651(05)70164-8. PMID 10986592